CLINICAL TRIAL: NCT02955745
Title: Plasma, Urine and Stools Appearance of an Orally Administered 129I-tracer for the Assessment of Dietary Iodine Absorption, Retention and Excretion in Humans: an Observational Study
Brief Title: Iodine-129 Tracer Method for Investigating Human Iodine Metabolism
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Swiss Federal Food Safety and Veterinary Office (Unknown); University Hospital, Zürich (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. dr. med., Swiss Federal Institute of Technology
Other Study IDs: Iodine-129
Record Dates: First submitted 2016-11-03; First posted 2016-11-04 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Iodine-129

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Other: Iodine-129 — The present study is an observational study and does not therefore include an investigational product in the proper sense because the used tracer (semi-stable iodine isotope) has no physiological effect on the participants. 129I will be used as tracer to measure appearance in plasma, urine and stools after the oral administered of the 129I-tracer.
  Other Names: 129I

SUMMARY:
Current iodine requirements defined for pregnancy and lactation are rough factorial estimates extrapolated from older studies in adults that used radioactive iodine tracers. To ensure optimal thyroid function in these vulnerable groups, a tracer method that could be safely used to accurately define iodine requirements would be valuable. Iodine-129 (129I), a long-lived semi-stable isotope with no health risks, could be used as a tracer, but the analytic challenges are formidable. However, we have developed an ICP-MS method to measure pp-billion (10-9) to pp-trillion (10-12) quantities of 129I in biological samples. In this project we will perform a study in which iodine-replete adult subjects will consume an oral dose of 129I. We will quantify 129I kinetic patterns in plasma, urine and stools after the oral dose, and use these data to derive tracer absorption, retention and excretion rates. This trial will allow us to define optimized procedures for the routine application of this method to assess iodine metabolism in humans. The use of 129I may prove to be a breakthrough technique to safely assess iodine metabolism and requirements in pregnant/lactating women in order to ensure healthy thyroid function in these age groups.

DETAILED DESCRIPTION:
Experimental design. The experimental design of this pilot-trial foresees the administration of a physiological oral dose of 12 µg of 129I (the tracer) in healthy adults coupled with quantitative measurement of the tracer concentration in plasma, urine, and stool samples collected prior and following tracer administration. A single dose of 12 µg 129I corresponds to a level of activity of 78.5 Bq and an exposure in adults of about 0.16 mSv for the thyroid as the target organ. Baseline plasma sample will be collected just before the administration of the tracer (-5 min) and follow-up samples will be collected 15, 30, 45, 60, and 90 min, as well as 2, 4, 8, 24, 48, 72, and 96 hours following tracer administration. Complete urine will be collected over a period of 8 days: baseline samples 1 day before the tracer dose (Day 3) and follow-up samples 7 days thereafter (until Day 10). Similarly, complete stool collection will be done on the day before the tracer dose (Day 3) as well as on the 3 following days (until Day 6). At Day 20 and 40 (follow-ups), blood sampling and spot urine collection will be repeated to verify washed out period. Baseline samples will be used for baseline-correction of post-administration samples. In order to minimize variability in the response for the purpose of this pilot-trial, the participants will consume a standardized diet during the first 6 days of the trial and will keep a food diary during the last 4 days of the trial. After suitable preparation, plasma, urine and stool samples will be analyzed for tracer quantification (determination of 129I mass on 127I mass; 127I being the naturally occurring iodine). From this data, we will construct pharmacokinetic curves of tracer appearance and clearance in blood, urine, and stool and we will derive rates and timing of human iodine absorption, retention and excretion. In addition, iodine speciation will be performed using iodine speciation based on a chromatography method coupled with ICP-MS for direct mass quantification of iodine species as plasma inorganic iodine (PII) and protein-bound iodine (PBI). This will provide an additional level of information on separate pharmacokinetics of metabolized and not metabolized 129I. Because uptake by the thyroid will be a determinant of the fraction of the tracer that is retained, the characterization of the participants' thyroid function is important to control for potential variation of calculated retention in our subjects, and thyroglobulin and thyroid hormones in whole blood will be assessed.

Methods of analysis. The tracer concentration in plasma, urine and stool will be measured by a high resolution multi collector ICP-MS with isotope dilution analysis (IDA) using a tellurium internal standard following sample digestion according to a method recently developed in our laboratory [Dold et al, Thyroid 2015]. For the additional speciation of 129I in plasma, analysis will be performed by using ion chromatography ICP-MS analysis (IC-ICP-MS) at the Federal Food Safety and Veterinary Office, Swizterland. Urinary iodine concentration will be measured by means of the Sandell-Kolthoff reaction [Pino et al, Clin Chem 1996, 42:239-243] in our laboratory. Thyroglobulin will be assessed using an ELISA dried blood spot method recently developed in our laboratory [Stinca et al, Thyroid 2015, 25:1297-1305]. Thyroid hormones will be measured by the University Hospital in Zurich, Switzerland, using a DELFIA (dissociation-enhanced lanthanide fluorescent immunoassay) method. Iodine content in the standardized diet will be will be measured in our laboratory by ICP-MS analysis and data from the food diaries will be evaluated by using the nutrition software EBIS-Pro (University of Hohenheim).

Data analysis and evaluation. The data generated by this pilot-trial will be used to construct pharmacokinetic curves of tracer appearance and clearance in the collected samples (total plasma, plasma PII-fraction, plasma PBI-fraction, urine, stools). Curves will be constructed by fitting a LOESS multiple regression model, a non-parametric locally weighted scatter plot smoothing of tracer concentration in samples as a function of time, and provide uncertainty range to visually represent the tracer's pharmacokinetic patterns and variability of response. For the evaluation of tracer kinetic patterns we will generate classic pharmacokinetic modelling parameters, including maximum tracer concentration (cmax), time at maximum tracer concentration (Tmax), elimination rate constant (ke), absorption rate constant (ka), and area under the curve (AUC), by using the simulation analysis and modelling software SAAM II (University of Washington). Total tracer retention will be calculated as total tracer intake - total tracer excreted (AUCurine + AUCstool). Total tracer absorption will be calculated as total tracer intake - total tracer appearance as plasma inorganic iodine (AUCPII). The optimization of procedures for routine application of this method will mainly include the definition of minimal requirements of specimen's specific sampling duration (number of days) after the administration of the tracer dose. This will be assessed by using ROC curves.

Expected output and significance/ expected impact. This study will be the first to use 129I as a biologic tracer in humans. Once developed, the availability of this novel method would provide a unique tool to address several key issues with regards to human iodine metabolism and thyroid function. These include the precise definition of the iodine requirement for important life stages, investigation of potential up-regulation of iodine absorption during iodine deficiency, thyroid uptake and turnover of iodine in varying iodine status, assessment of placental and breast milk iodine transfer, as well as the assessment of iodine bioavailability from different foods. Thus, this project could have significant long term impact in the field of iodine and the thyroid.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 45 years
2. Body weight <80 kg and BMI 19-27.5
3. Current use of iodized salt at home
4. Signed informed consent
5. Good knowledge of English language

Exclusion Criteria:

1. Inadequate iodine status (defined as UIC <80 µg/L or >300 µg/L and assessed during screening from 10 urine spot samples)
2. Exposure to iodine-containing X-ray/ computed tomography contrast agent
3. Use of iodine-containing disinfectants (betadine)
4. History of thyroid disease (according to the participants own statement)
5. Any metabolic, gastrointestinal or chronic disease such as diabetes, hepatitis, hypertension, or cancer (according to the participants own statement)
6. Chronic use of medications (except for contraceptives)
7. Use of iodine containing supplements within 6 months prior to study start
8. Pregnancy (according to the participants own statement but confirmed by a pregnancy test with the first urine spot sample from screening)
9. Breast feeding
10. Vegan or vegetarian diet
11. Drug abuse
12. Extensive alcohol intake, defined as more than 3 (men) or 2 (women) standard drinks per day (i.e. 3dl beer, 1dl wine, 3-4cl liquor), with less than 2 days per week without alcohol consumption
13. Earlier participation in any other clinical study within the last 30 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Generally healthy, iodine-replete males and non-pregnant, non-lactating females, who are between 18 and 45 years old, whose body weight is less than 80 kg and BMI between 19-27.5 kg/m2, who regularly consume iodized salt, who have signed the informed consent, and who have good knowledge of the English language. They will serve as an iodine-sufficient population with normal iodine metabolism.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-11; Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
129I kinetics | 8 days
  129I-tracer concentration in plasma (both in its inorganic and organic form), urine, and stool samples collected prior and following administration of a single physiological oral 129I dose in order to derive rates of absorption, retention, and excretion of dietary iodine

SECONDARY OUTCOMES:
Thyroid function | 1 day
  Quantitative assessment of participants' thyroglobulin and thyroid hormones in circulation (thyroid function tests)
Dietary iodine | 10 days
  Quantitative assessment of iodine content in the participants' diet
Minimal sampling requirements | 10 days
  Definition of the minimal requirements of specimen's specific sampling duration (number of days) after the administration of the 129I dose

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, MD, Principal Investigator — ETH Zurich
Locations (1):
- ETH Zurich, Laboratory of Human Nutrition, Zurich, Switzerland